CLINICAL TRIAL: NCT03263728
Title: Cardiac Magnetic Resonance for Asymptomatic Type 2 Diabetics With Cardiovascular High Risk (CATCH) - Pilot Study
Acronym: CATCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Radiological Society of North America (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UW-17-168
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus, Type 2; Coronary Artery Disease
Keywords: Stress Cardiac Magnetic Resonance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stress Cardiac MR (Experimental)
  Interventions: Diagnostic Test: Cardiac Magnetic Resonance

INTERVENTIONS:
Diagnostic Test: Cardiac Magnetic Resonance — Screening of asymptomatic of high risk type 2 diabetic mellitus patients with stress cardiac magnetic resonance

SUMMARY:
The aim of this study is to determine the prevalence of myocardial ischaemia in asymptomatic high risk type 2 diabetic patients using stress cardiac MR and how many stress cardiac MR examinations are false positive.

DETAILED DESCRIPTION:
Asymptomatic coronary artery disease (CAD) is highly prevalent (ie. 17-59%) in type 2 diabetic patients. In addition, cardiovascular disease remains the most common cause of death in type 2 diabetics. Previous trials using coronary computed tomography angiograms (CCTA) or nuclear myocardial perfusion imaging (MPI) to screen for asymptomatic coronary artery disease requiring intervention have been unsuccessful at reducing cardiovascular and all cause mortality when compared to optimised medical therapy where cardiovascular risk factors are treated in order to reduce cardiovascular complications. Possible reasons for this include, the choice of imaging modality, the intervention chosen (eg. bare metal stents vs drug eluting stents), patient cohort (eg. all diabetics vs high risk diabetics). Stress cardiac magnetic resonance (CMR) is ideally suited to assess this group of high risk patients as there is no radiation exposure and it allows a more complete analysis of the heart including the assessment of myocardial viability, cardiac systolic and diastolic function. The significance of this envisioned randomised controlled trial is firstly to investigate if stress CMR screening will reduce major adverse cardiovascular events including death. Secondly, a study using stress CMR has never been performed.

ELIGIBILITY:
Inclusion Criteria:

* Onset of type 2 diabetes at ≥30yrs old with no history of ketoacidosis
* 60-80yrs old
* Framingham Risk Score ≥20%

Exclusion Criteria:

* Angina pectoris or chest discomfort
* Stress test or coronary angiography within 2 years
* Previous myocardial infarction (MI)
* Previous coronary artery stenting or coronary artery bypass grafting
* Any clinical indication or contraindication for stress testing
* Any contraindication to stress CMR (eg. non-MRI compatible devices)
* Contraindication to gadolinium based contrast agent (eg. Renal impairment with an estimated glomerular filtration rate (GFR) <30ml/min/1.73m2)
* Life expectancy <2 years due to cancer or liver disease
* Contraindication to dual antiplatelet therapy
* Planned need for concomitant cardiac surgery
* Refusal or inability to sign an informed consent.
* Potential for non-compliance towards the requirements in the trial protocol
* Unable to cover the costs of percutaneous coronary intervention (PCI) whether through government subsidies, etc

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-01-29 (Actual)

PRIMARY OUTCOMES:
Prevalence of myocardial ischaemia | 1 year

SECONDARY OUTCOMES:
Prevalence of myocardial infarction | 1 year
Clinical predictors of silent ischaemia | 1 year
Major adverse cardiovascular events | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Ng MY, Zhou W, Vardhanabhuti V, Lee CH, Yu EYT, Wan EYF, Chan K, Yan AT, Ip TP, Yiu KH, Wintersperger BJ. Cardiac magnetic resonance for asymptomatic patients with type 2 diabetes and cardiovascular high risk (CATCH): a pilot study. Cardiovasc Diabetol. 2020 Mar 31;19(1):42. doi: 10.1186/s12933-020-01019-2. PMID 32234045